CLINICAL TRIAL: NCT04421482
Title: Cold Milk as a Novel Therapy for Dysphagia in Preterm Infants
Brief Title: Cold Milk for Dysphagia in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-00876; R21HD100653 (NIH)
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Dysphagia of Newborn
MeSH Terms: interventions — Cold Temperature

STUDY DESIGN:
Intervention Model Description: This will be a prospective study, with each infant serving as their own control. The order of each condition will be randomized to control for fatigue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Very Low Birth Weight Preterm Infants (Other): Very Low Birth Weight Preterm Infants (birth weight less than 1,500g and less than 32 weeks gestation) admitted to NYU Winthrop NICU. Infants will first receive room temperature milk and then be assessed for signs of dysphagia. Only infants that show signs of dysphagia will receive cold milk.
  Interventions: Other: Standard room temperature (RTS) feeding of milk/formula; Other: Cold temperature (CS, at 4-9°C) of milk/formula

INTERVENTIONS:
Other: Standard room temperature (RTS) feeding of milk/formula — Standard room temperature (RTS) milk/formula will be given for an entire feeding (15-20 minutes).
Other: Cold temperature (CS, at 4-9°C) of milk/formula — If the infant shows signs of dysphagia cold temperature (CS, at 4-9°C) milk/formula will be given for an entire feeding (15-20 minutes).

SUMMARY:
It is estimated that 30-70% of very low birth weight (VLBW) preterm infants will be diagnosed with swallowing dysfunction (dysphagia), which often leads to airway compromise in the form of laryngeal penetration and/or tracheal aspiration during oral feeding attempts. Chronic airway compromise results in a persistent inflammatory state, with disease progression that can be devastating for already fragile and developmentally immature lungs in preterm infants. At this time, there are limited therapeutic options for dysphagia in VLBW infants during oral feeding. In a recent publication, our research group was the first to demonstrate that short-duration of oral feeding with cold liquid reduces dysphagia occurrence from 71% to 26%. However, these data must be further validated for the effectiveness and safety of a full duration feeding before being recommended for routine clinical practice.

The objective is to identify preliminary evidence for the efficacy and safety of feeding full oral cold milk for dysphagia management in preterm infants. We hypothesize that oral feeding of cold milk in VLBW preterm infants with dysphagia will improve suck/swallow/breathe coordination and decrease penetration/ aspiration to the airway. We further hypothesize that cold milk intervention will have no adverse effects on intestinal blood flow, as assessed by Doppler Ultrasound. This is significant because there is a critical need to identify effective and safe evidence-based treatment options for dysphagia management in preterm infants.

This prospective study will seek to enroll Subjects who meet the following inclusion criteria: 1) VLBW (birth weight less than 1,500g and less than 32 weeks gestation), 2) admitted to NYU-Winthrop Neonatal Intensive Care Unit (NICU), 3) Post-menstrual age (PMA) > 35 weeks at the time of the study, 4) receiving no or minimum respiratory support (<1 lit/min low-flow nasal cannula), 5) tolerating at least 50% of their enteral feeding orally, 6) having symptoms of swallowing dysfunction during oral feeding (clinical dysphagia) and 7) referred by the medical team for video fluoroscopic swallow study (VFSS) and/or fiberoptic endoscopic evaluation of swallowing (FEES).

To assess the efficacy of cold milk in treating dysphagia, study subjects will first have an oral motor feeding assessment using an FDA approved device called the nFant® Feeding Solution as well as VFSS and/or FEES. To assess the safety of using cold milk, subjects will receive a doppler ultrasound before and after the ingestion of cold liquid feeding to assess the mesenteric blood flow.

ELIGIBILITY:
Inclusion Criteria:

1. Viable preterm infants less than 34 weeks gestation
2. admitted to NYU- Langone Long Island Hospital NICU
3. PMA > 35 weeks at the time of the study
4. receiving no or minimum respiratory support (<2 lit/min low-flow nasal cannula)
5. tolerating at least 50% of their enteral feeding orally and
6. having symptoms of swallowing dysfunction during oral feeding (clinical dysphagia).
7. referred by the medical team for VFSS and/or FEES assessments.

Exclusion Criteria:

Infants with other comorbidities, such as IUGR, upper airway anomalies, brain injury, neuromuscular disease, or life-threatening congenital disease.

Min Age: 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nazeeh Hanna, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Nazeeh.hanna@NYULangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Researchers who provide a methodologically sound proposal may direct requests to Nazeeh.hanna@NYULangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Ferrara-Gonzalez L, Kamity R, Htun Z, Dumpa V, Islam S, Hanna N. From Warm to Cold: Feeding Cold Milk to Preterm Infants with Uncoordinated Oral Feeding Patterns. Nutrients. 2025 Apr 26;17(9):1457. doi: 10.3390/nu17091457. PMID 40362766
- [Derived] Ferrara L, Kamity R, Htun Z, Dumpa V, Islam S, Hanna N. From Warm to Cold: Feeding Cold Milk in Preterm Infants with Uncoordinated Oral Feeding Patterns. Res Sq [Preprint]. 2024 Jun 18:rs.3.rs-4504972. doi: 10.21203/rs.3.rs-4504972/v1. PMID 38947097

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Very Low Birth Weight Preterm Infants
Started | 22
Completed | 21
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Very Low Birth Weight Preterm Infants
Number analyzed (Participants) | 21
Age, Continuous [Median (Inter-Quartile Range); unit: weeks gestation] | 32 [28 to 33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 12
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Infants With Improvement of Dysphagia
Description: Dysphagia will be assessed by Video Fluoroscopic Swallow Study (VFSS) and/or Fiberoptic Endoscopic Evaluation of Swallowing (FEES). If the infants showed signs of dysphagia they would receive cold cold milk and improvements in dysphagia would be assessed again by VFSS and FEES.
Time Frame: 15-20 minutes post cold milk feeding
Population: Infants were assessed post room temp milk feeding for dysphagia. If they showed signs of dysphagia, they would receive cold milk. Therefore only infants showing dysphagia either by FEES or VFSS were included in the analysis, as not all infants received cold milk during this assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Very Low Birth Weight Preterm Infants
Number analyzed (Participants) | 12
Percentage of patients | 58 [30.4 to 86.3]

2. Primary Outcome: Axillary Temperature of Infants Post Room Temperature Feeding
Description: Outcome measure will be assessed by measuring Axillary temperatures. The axillary temperature will be taken directly after feeding.
Time Frame: Post feeding (up to 5 minutes)
Measure: Mean (Standard Deviation); unit: Degrees fahrenheit
Groups:
- Standard Room Temperature (RTS) Feeding of Milk/Formula (Control): Very Low Birth Weight Preterm Infants (birth weight less than 1,500g and less than 32 weeks gestation) admitted to NYU Winthrop NICU. Infants will first receive room temperature milk and then be assessed for signs of dysphagia. Only infants that show signs of dysphagia will receive cold milk.
Arm/Group | Standard Room Temperature (RTS) Feeding of Milk/Formula (Control)
Number analyzed (Participants) | 21
Degrees fahrenheit | 98.2 (0.3)

3. Primary Outcome: Percentage of Infants With Change in Vital Signs Due to Cold Milk
Description: Outcome measure will be assessed by monitoring changes in respiratory rate, heart rate, and oxygen saturation.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Very Low Birth Weight Preterm Infants
Number analyzed (Participants) | 12
Participants | 0

4. Primary Outcome: Change in Peak Systolic Velocity (PSV) (60 Minutes Post Feeding)
Description: Outcome measure will be assessed by abdominal ultrasound. Peak systolic velocity (PSV) was measured for each patient before feeding (room temp or cold milk) as well as 60 minutes after feeding (room temp and cold milk).
Time Frame: Baseline (prior to feeding), 60 minutes after feeding
Population: The outcome measure was not collected after the first five infants, as the analysis showed no significant change. As a result, there was no justification for continuing data collection or subjecting the remaining infants to the procedure.
Measure: Mean (95% Confidence Interval); unit: cm/s
Arm/Group | Very Low Birth Weight Preterm Infants
Number analyzed (Participants) | 5
cm/s | 1.1 [-10 to 12.3]

ADVERSE EVENTS:
Time Frame: 60 minutes
Description: Study team members were responsible for documenting any side effect by direct assessment and observation.
Arm/Group | Very Low Birth Weight Preterm Infants
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/82/NCT04421482/Prot_SAP_001.pdf
  • Informed Consent Form (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/82/NCT04421482/ICF_000.pdf